CLINICAL TRIAL: NCT06842758
Title: Relationship Between Thoracic Hyperkyphosis and Fall Risk in Women with Fragility Vertebral Fractures
Status: Active, not recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Other Study IDs: MFR012025
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis; Hyperkyphosis; Vertebral Body Fracture
Keywords: osteoporosis; Hyperkyphosis; vertebral body fracture; rehabilitation
MeSH Terms: conditions — Osteoporosis; Kyphosis | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: A group of 18 women aged ≥65 years with the presence of at least three documented vertebral fragility fractures and diagnosis of thoracic hyperkyphosis.
  Interventions: Other: Rehabilitation Treatment
- Group B: A group of 22 women aged ≥65 years with the presence of at least three documented vertebral fragility fractures and diagnosis of thoracic hyperkyphosis.
  Interventions: Other: None Treatment

INTERVENTIONS:
Other: Rehabilitation Treatment — Group A patients came to our department to perform rehabilitation treatment. They underwent rehabilitation treatment for a total of 20 rehabilitation sessions, performed on a daily basis lasting 60 minutes, on a 1:1 basis with a physical therapist, . They performed postural re-education and posterior kinetic chain strengthening exercises.
  Groups: Group A
Other: None Treatment — Group B patients did not undergo rehabilitation treatment. They underwent subcutaneous Teriparatide drug treatment on a daily basis for the treatment of osteoporosis
  Groups: Group B

SUMMARY:
Multiple vertebral fragility fractures, one of the main complications of osteoporosis, are frequently associated with thoracic hyperkyphosis, which in turn leads to significant postural alterations.

These biomechanical changes may increase fall risk, posing a critical clinical issue for elderly patients. However, the results of studies investigating the association between hyperkyphosis and fall risk are conflicting, highlighting the need for further research.

This study aims to explore the correlation between the severity of thoracic kyphotic curvature and fall risk in patients with multiple fragility fractures undergoing osteoporosis treatment.

Additionally, the study seeks to evaluate the role of physiotherapy in improving patients' functional and postural outcomes.

A retrospective observational study was conducted, supplemented by a narrative literature review to contextualize the findings. Forty patients undergoing treatment at the Functional Recovery and Rehabilitation Unit (UOC) of P. Giaccone University Hospital in Palermo were enrolled and followed up via biannual phone interviews. Data were collected between May 2023 and May 2024, with a longitudinal assessment of outcomes from T0 (baseline) to T1 (12 months).

The severity of the kyphotic curve was quantified using the Cobb method, while fall risk was assessed through the Berg Balance Scale. Participation in physiotherapy programs was analyzed to evaluate their impact on clinical and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥65 years.
* Presence of at least three documented vertebral fragility fractures.
* Diagnosis of thoracic hyperkyphosis

Exclusion Criteria:

* History of orthopedic surgeries involving the spine or lower limbs.
* Treatments for cerebrovascular diseases.
* Presence of balance disorders.
* Active oncological diseases.
* Use of walking aids

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: A group of 40 women aged ≥65 years with the presence of at least three documented vertebral fragility fractures and a diagnosis of thoracic hyperclyphosis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Degree of Hyperkyphosis | At the baseline specialist assessment (T0); After one year from the baseline specialist assessment (T1);
  Cobb's method by 2p radiographic examination of the whole spine
Number of falls in the last year | At the baseline specialist assessment (T0); After one year from the baseline specialist assessment (T1);
  Evaluation of the number of falls in the last year
Balance | At the baseline specialist assessment (T0); After one year from the baseline specialist assessment (T1);
  Assessment of balance by means of the Berg Scale

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. P. Giaccone, Palermo, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Scaturro D, Rizzo S, Sanfilippo V, Giustino V, Messina G, Martines F, Falco V, Cuntrera D, Moretti A, Iolascon G, Letizia Mauro G. Effectiveness of Rehabilitative Intervention on Pain, Postural Balance, and Quality of Life in Women with Multiple Vertebral Fragility Fractures: A Prospective Cohort Study. J Funct Morphol Kinesiol. 2021 Mar 3;6(1):24. doi: 10.3390/jfmk6010024. PMID 33802536
- [Background] Tarantino U, Iolascon G, Cianferotti L, Masi L, Marcucci G, Giusti F, Marini F, Parri S, Feola M, Rao C, Piccirilli E, Zanetti EB, Cittadini N, Alvaro R, Moretti A, Calafiore D, Toro G, Gimigliano F, Resmini G, Brandi ML. Clinical guidelines for the prevention and treatment of osteoporosis: summary statements and recommendations from the Italian Society for Orthopaedics and Traumatology. J Orthop Traumatol. 2017 Nov;18(Suppl 1):3-36. doi: 10.1007/s10195-017-0474-7. PMID 29058226
- [Background] Cultrera P, Pratelli E, Petrai V, Postiglione M, Zambelan G, Pasquetti P. Evaluation with stabilometric platform of balance disorders in osteoporosis patients. A proposal for a diagnostic protocol. Clin Cases Miner Bone Metab. 2010 May;7(2):123-5. PMID 22460016